CLINICAL TRIAL: NCT02225340
Title: Relationships Between Plasma PCSK9 Levels, LDL-cholesterol Concentrations and Lipoprotein (a) Levels in Familial Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Couture, MD, FRCP, PhD, Laval University
Other Study IDs: FH-PCSK9
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls
- Familial hypercholesterolemia

SUMMARY:
Familial hypercholesterolemia (FH) is an autosomal codominant single gene disorder caused by mutations in the LDL receptor gene (LDLR) that disrupt the normal clearance of LDL particles from the plasma. Heterozygous patients (HeFH) present a two- to three-fold raise in plasma LDL-cholesterol (LDL-C) concentrations and coronary artery disease occurs earlier among HeFH carrying negative-receptor (NR) mutations as compared with HeFH subjects carrying defective-receptor (DR) variants. Proprotein convertase subtilisin/kexin type 9 (PCSK9) regulates LDL-C levels by binding to LDLR and by enhancing its intracellular degradation.

The objective of this study is to examine to what extent variations in LDL-C and Lipoprotein (Lp) (a) concentrations are related to PCSK9 levels in a large French-Canadian cohort of HeFH subjects.

The primary hypothesis is that that PCSK9 levels have a significant impact on LDL-C concentration variability and are associated with Lp(a) levels.

ELIGIBILITY:
Inclusion Criteria:

Subjects with familial hypercholesterolemia:

* Aged between 18-65 years
* Carrier of a mutation in the LDL receptor gene

Controls:

* Aged between 18-60 years
* HDL-cholesterol > 1.1 mmol/L
* Triglycerides < 1.7 mmol/L
* Fasting blood glucose <6.1 mmol/L
* Normal blood pressure (<130/85)

Exclusion Criteria:

* Subjects with a previous history of cardiovascular disease
* Subjects with Type 2 diabetes
* Were pregnant or nursing;
* Subjects with a history of cancer
* Subjects with acute liver disease, hepatic dysfunction, or persistent elevations of serum transaminases
* Subjects with a secondary hyperlipidemia due to any cause
* History of alcohol or drug abuse within the past 2 years
* hormonal treatment
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Impact of PCSK9 on LDL-C concentrations | Week 1

SECONDARY OUTCOMES:
Impact of PCSK9 on Lp(a) concentrations | Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, FRCP, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada

REFERENCES:
- [Derived] Drouin-Chartier JP, Hogue JC, Tremblay AJ, Bergeron J, Lamarche B, Couture P. The elevation of plasma concentrations of apoB-48-containing lipoproteins in familial hypercholesterolemia is independent of PCSK9 levels. Lipids Health Dis. 2017 Jun 15;16(1):119. doi: 10.1186/s12944-017-0502-x. PMID 28619117